CLINICAL TRIAL: NCT03550313
Title: A PHASE 2, RANDOMIZED, OPEN-LABEL TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF A MULTIVALENT PNEUMOCOCCAL CONJUGATE VACCINE GIVEN WITH, OR SEPARATELY FROM, 13-VALENT PNEUMOCOCCAL CONJUGATE VACCINE IN HEALTHY INFANTS
Brief Title: Study to Evaluate the Safety and Immunogenicity of a Multivalent Pneumococcal Vaccine Given With Prevnar 13 in Healthy Infants
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study vaccinations and blood draws were halted due to adequacy of a smaller dataset and study feasibility issues. It was not based on any safety concerns.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C3571002; 2020-005039-59 (EudraCT Number)
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Results first posted 2021-11-30 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — Vaccines, Combined; Pneumococcal Vaccines; 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1 - Coadministration (Experimental): Multivalent pneumococcal conjugate vaccine coadministered with Prevnar 13
  Interventions: Biological: Multivalent; Biological: Prevnar 13
- Group 2 - Staggered Administration (Experimental): Multivalent pneumococcal conjugate vaccine given 1 month after Prevnar 13
  Interventions: Biological: Multivalent; Biological: Prevnar 13
- Group 3 - Control with Supplemental Dose (Active Comparator): Prevnar 13 with a single dose of multivalent pneumococcal conjugate vaccine
  Interventions: Biological: Multivalent; Biological: Prevnar 13

INTERVENTIONS:
Biological: Multivalent — Pneumococcal conjugate vaccine
  Other Names: Pneumococcal conjugate vaccine
Biological: Prevnar 13 — Pneumococcal conjugate vaccine

SUMMARY:
This is a Phase 2, randomized, active-controlled, open-label study with a 3-arm parallel design. Healthy 2-month old infants (42 to 98 days of age) with no history of pneumococcal vaccination will be randomized in a 1:1:1 ratio to receive a 4-dose series of: multivalent pneumococcal conjugate vaccine coadministered with Prevnar 13 (Group 1); multivalent pneumococcal conjugate vaccine given 1 month after Prevnar 13 (Group 2); or Prevnar 13 with a single dose of multivalent pneumococcal conjugate vaccine (Group 3).

ELIGIBILITY:
Inclusion Criteria:

* Male or female infant born at >36 weeks of gestation and aged 2 months (42 to 98 days) at the time of consent (the day of birth is considered day of life 1).
* Healthy infant determined by medical history, physical examination, and clinical judgment.

Exclusion Criteria:

* Previous vaccination with licensed or investigational pneumococcal vaccine.
* Prior receipt of routine pediatric vaccines, with the exception of hepatitis B vaccine.
* Previous receipt of >1 dose of hepatitis B vaccine.
* Prior hepatitis B vaccine must have been administered at age <30 days.
* Major known congenital malformation or serious chronic disorder.
* Receipt of blood/plasma products or immunoglobulins.

Ages: 42 Days to 98 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 565 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (48):
- United States (48):
  - Mobile Pediatric Clinic, Mobile, Alabama
  - Harrisburg Family Medical Center, Harrisburg, Arkansas
  - Emmaus Research Center, Inc., Anaheim, California
  - Hoag Memorial Hospital Presbyterian, Huntington Beach, California
  - Madera Family Medical Group, Madera, California
  - Orange County Research Institute, Ontario, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Center for Clinical Trials, Paramount, California
  - Gentle Medicine Associates, Boynton Beach, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Next Phase Research Alliance, Homestead, Florida
  - Acevedo Clinical Research Associates, Miami, Florida
  - Bio-Medical Research, LLC, Miami, Florida
  - Crystal Biomedical Research, LLC, Miami Lakes, Florida
  - IACT Health, Columbus, Georgia
  - Advocate Children's Hospital, Park Ridge, Illinois
  - MOC Research, Mishawaka, Indiana
  - Michael W. Simon, MD, PSC, Lexington, Kentucky
  - All Children Pediatrics, Louisville, Kentucky
  - Meridian Clinical Research, LLC, Baton Rouge, Louisiana
  - MedPharmics, LLC, Metairie, Louisiana
  - LSUHSC-Shreveport, Shreveport, Louisiana
  - Ochsner-LSU Health Shreveport, Shreveport, Louisiana
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - Pediatric Phlebotomy, Boston, Massachusetts
  - Tufts Medical Center IDS - Pharmacy, Boston, Massachusetts
  - Children's Mercy Clinics on Broadway, Kansas City, Missouri
  - Children's Physicians Embassy Park, Omaha, Nebraska
  - Children's Physicians Spring Valley, Omaha, Nebraska
  - Creighton University Clinical Research Office, Omaha, Nebraska
  - Child Health care Associates, East Syracuse, New York
  - Blue Ridge Pediatric and Adolescent Medicine, Inc, Boone, North Carolina
  - Sugarcamp Family Research, Dayton, Ohio
  - Allegheny Health and Wellness Pavilion, Erie, Pennsylvania
  - Coastal Pediatric Research, Charleston, South Carolina
  - Parkside Pediatrics, Greenville, South Carolina
  - Sanford Children's Specialty Clinic, Sioux Falls, South Dakota
  - Sanford Research, Sioux Falls, South Dakota
  - Sanford 69th & Louise Family Medicine, Sioux Falls, South Dakota
  - Holston Medical Group, Kingsport, Tennessee
  - Ventavia Research Group, Houston, Texas
  - Mercury Clinical Research, Houston, Texas
  - Pediatric Associates, Houston, Texas
  - Ventavia Research Group, Keller, Texas
  - Tekton Research, Inc., San Antonio, Texas
  - Ventavia Research Group, LLC, Spring, Texas
  - Dixie Pediatrics, St. George, Utah
  - Marshall Health, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Simon MW, Bataille R, Caldwell NS, Gessner BD, Jodar L, Lamberth E, Peng Y, Scott DA, Lei L, Giardina PC, Gruber WC, Jansen KU, Thompson A, Watson W. Safety and immunogenicity of a multivalent pneumococcal conjugate vaccine given with 13-valent pneumococcal conjugate vaccine in healthy infants: A phase 2 randomized trial. Hum Vaccin Immunother. 2023 Aug;19(2):2245727. doi: 10.1080/21645515.2023.2245727. Epub 2023 Nov 5. PMID 37927075
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3571002

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 569 infants had a signed informed consent document; 4 of these infants were deemed ineligible before randomization, and did not participate further. 565 participants were randomized in 3 reporting groups- 512 participants from 39 sites and 53 from 2 terminated sites (terminated due to serious quality issues). The study includes and reports valid data only from 512 participants. Out of these 512 participants, 484 received at least 1 vaccination.
Groups:
- Group 1: c7vPnC and Prevnar 13 Co-administration: Participants who received a dose of complementary 7-valent pneumococcal conjugate vaccine (c7vPnC) in one leg at 2, 4, 6 and 12 months of age (Dose 1, 2, 3, and 4 respectively) and Prevnar 13 at 2, 4, 6, and 12 months of age in another leg.
- Group 2: c7vPnC and Prevnar 13 Staggered Administration: Participants who received a dose of c7vPnC at 3, 5, 7, and 13 months of age in one leg (Dose 1, 2, 3, and 4 respectively) and Prevnar 13 at 2, 4, 6, and 12 month of age in another leg.
- Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose: Participants who received a dose of Prevnar 13 at 2, 4, 6, and 12 months of age (Dose 1, 2, 3, and 4 respectively) and a dose of c7vPnC at 13 months of age (Supplemental Dose).
Period: Overall Study
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Started | 192 | 187 | 186
Vaccinated for Dose 1 | 171 | 147 | 166
Vaccinated for Dose 2 | 159 | 135 | 153
Vaccinated for Dose 3 | 151 | 127 | 146
Completed | 95 | 77 | 72
Not Completed | 97 | 110 | 114
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Lost to Follow-up | 5 | 7 | 12
Not completed — Study terminated by sponsor | 44 | 37 | 48
Not completed — No longer met eligibility criteria | 3 | 5 | 6
Not completed — Withdrawal by parent/guardian | 20 | 18 | 26
Not completed — Other | 4 | 2 | 2
Not completed — Randomized but not vaccinated | 3 | 23 | 2
Not completed — Sites terminated due to quality issues | 18 | 17 | 18

BASELINE CHARACTERISTICS:
Population: The overall safety population included all participants who received at least 1 dose of c7vPnC (in Groups 1 and 2) or Prevnar 13 (in Group 3) and had safety data reported in the study.
Groups:
- Group 1: c7vPnC and Prevnar 13 Co-administration: Participants who received a dose of c7vPnC in one leg at 2, 4, 6 and 12 months of age (Dose 1, 2, 3, and 4 respectively) and Prevnar 13 at 2, 4, 6, and 12 months of age in another leg.
- Total: Total of all reporting groups
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose | Total
Number analyzed (Participants) | 171 | 147 | 166 | 484
Age, Continuous [Mean (Standard Deviation); unit: Days] | 65.9 (9.53) | 95.1 (10.40) | 64.9 (8.22) | 74.4 (16.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 80 | 75 | 240
  Male | 86 | 67 | 91 | 244
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 89 | 70 | 85 | 244
  Not Hispanic or Latino | 81 | 77 | 80 | 238
  Unknown or Not Reported | 1 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 8 | 3 | 15
  Asian | 7 | 5 | 3 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 35 | 26 | 31 | 92
  White | 102 | 90 | 105 | 297
  More than one race | 6 | 4 | 6 | 16
  Unknown or Not Reported | 17 | 14 | 17 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 1
Description: Local reactions were recorded using an electronic diary (e-diary) by participant's legally acceptable representative (LAR). Local reactions included redness, swelling and pain at the injection site. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 centimeter (cm). Redness and swelling were graded as mild (greater than [>] 0.0 to 2.0 cm), moderate (>2.0 to 7.0 cm) and severe (>7 cm). Pain at injection site was graded as mild (hurt if gently touched), moderate (hurt if gently touched, with crying), and severe (caused limitation of limb movement).
Time Frame: Within 7 Days After Dose 1
Population: The overall safety population included all participants who received at least 1 dose of c7vPnC (in Groups 1and 2) or Prevnar 13 (in Group 3) and had safety data reported in the study. Here, "Overall Number of Participants Analyzed" signifies number of participants with any e-diary data reported after Dose 1 in the overall safety population. Dose 1 was first dose of c7vPnC in Group 1 and Group 2, and first dose of Prevnar 13 in Group 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 166 | 144 | 165
Percentage of participants
  Redness: Any | 25.9 [19.4 to 33.3] | 26.4 [19.4 to 34.4] | 21.8 [15.8 to 28.9]
  Redness: Mild | 16.3 [11.0 to 22.8] | 21.5 [15.1 to 29.1] | 18.2 [12.6 to 24.9]
  Redness: Moderate | 9.6 [5.6 to 15.2] | 4.9 [2.0 to 9.8] | 3.6 [1.3 to 7.7]
  Redness: Severe | 0 [0.0 to 2.2] | 0 [0.0 to 2.5] | 0 [0.0 to 2.2]
  Swelling: Any | 27.1 [20.5 to 34.5] | 22.2 [15.7 to 29.9] | 23.6 [17.4 to 30.9]
  Swelling: Mild | 16.3 [11.0 to 22.8] | 13.9 [8.7 to 20.6] | 17.0 [11.6 to 23.6]
  Swelling: Moderate | 10.2 [6.1 to 15.9] | 8.3 [4.4 to 14.1] | 5.5 [2.5 to 10.1]
  Swelling: Severe | 0.6 [0.0 to 3.3] | 0 [0.0 to 2.5] | 1.2 [0.1 to 4.3]
  Pain at Injection Site: Any | 59.6 [51.8 to 67.2] | 40.3 [32.2 to 48.8] | 50.3 [42.4 to 58.2]
  Pain at Injection Site: Mild | 28.9 [22.2 to 36.4] | 28.5 [21.3 to 36.6] | 26.1 [19.5 to 33.5]
  Pain at Injection Site: Moderate | 27.7 [21.1 to 35.2] | 11.1 [6.5 to 17.4] | 22.4 [16.3 to 29.6]
  Pain at Injection Site: Severe | 3.0 [1.0 to 6.9] | 0.7 [0.0 to 3.8] | 1.8 [0.4 to 5.2]

2. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 2
Description: Local reactions were recorded using an electronic diary by participant's LAR. Local reactions included redness, swelling and pain at the injection site. Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit =0.5 cm. Redness and swelling were graded as mild (>0.0 to 2.0 cm), moderate (>2.0 to 7.0 cm) and severe (>7 cm). Pain at injection site was graded as mild (hurt if gently touched), moderate (hurt if gently touched, with crying), and severe (caused limitation of limb movement).
Time Frame: Within 7 Days After Dose 2
Population: The overall safety population included all participants who received at least 1 dose of c7vPnC (in Groups 1 and 2) or Prevnar 13 (in Group 3) and had safety data reported in the study. Here, "Overall Number of Participants Analyzed" signifies number of participants with any e-diary data reported after vaccination in the overall safety population. Dose 2 was second dose of c7vPnC in Group 1 and Group 2, and second dose of Prevnar 13 in Group 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 152 | 126 | 147
Percentage of participants
  Redness: Any | 28.9 [21.9 to 36.8] | 20.6 [13.9 to 28.8] | 23.8 [17.2 to 31.5]
  Redness: Mild | 22.4 [16.0 to 29.8] | 18.3 [11.9 to 26.1] | 21.1 [14.8 to 28.6]
  Redness: Moderate | 6.6 [3.2 to 11.8] | 2.4 [0.5 to 6.8] | 2.7 [0.7 to 6.8]
  Redness: Severe | 0 [0.0 to 2.4] | 0 [0.0 to 2.9] | 0 [0.0 to 2.5]
  Swelling: Any | 21.1 [14.9 to 28.4] | 16.7 [10.6 to 24.3] | 22.4 [16.0 to 30.1]
  Swelling: Mild | 14.5 [9.3 to 21.1] | 14.3 [8.7 to 21.6] | 16.3 [10.7 to 23.3]
  Swelling: Moderate | 6.6 [3.2 to 11.8] | 2.4 [0.5 to 6.8] | 6.1 [2.8 to 11.3]
  Swelling: Severe | 0 [0.0 to 2.4] | 0 [0.0 to 2.9] | 0 [0.0 to 2.5]
  Pain at Injection Site: Any | 55.3 [47.0 to 63.3] | 23.8 [16.7 to 32.2] | 46.9 [38.7 to 55.3]
  Pain at Injection Site: Mild | 31.6 [24.3 to 39.6] | 19.0 [12.6 to 27.0] | 27.9 [20.8 to 35.9]
  Pain at Injection Site: Moderate | 21.7 [15.4 to 29.1] | 4.8 [1.8 to 10.1] | 18.4 [12.5 to 25.6]
  Pain at Injection Site: Severe | 2.0 [0.4 to 5.7] | 0 [0.0 to 2.9] | 0.7 [0.0 to 3.7]

3. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 3
Description: as for outcome 2
Time Frame: Within 7 Days After Dose 3
Population: The overall safety population included all participants who received at least 1 dose of c7vPnC (in Groups 1 and 2) or Prevnar 13 (in Group 3) and had safety data reported in the study. Here, "Overall Number of Participants Analyzed" signifies number of participants with any e-diary data reported after vaccination in the overall safety population. Dose 3 was third dose of c7vPnC in Group 1 and Group 2, and third dose of Prevnar 13 in Group 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 143 | 120 | 138
Percentage of participants
  Redness: Any | 25.2 [18.3 to 33.1] | 20.0 [13.3 to 28.3] | 22.5 [15.8 to 30.3]
  Redness: Mild | 23.1 [16.4 to 30.9] | 19.2 [12.6 to 27.4] | 18.1 [12.1 to 25.6]
  Redness: Moderate | 2.1 [0.4 to 6.0] | 0.8 [0.0 to 4.6] | 4.3 [1.6 to 9.2]
  Redness: Severe | 0 [0.0 to 2.5] | 0 [0.0 to 3.0] | 0 [0.0 to 2.6]
  Swelling: Any | 21.7 [15.2 to 29.3] | 14.2 [8.5 to 21.7] | 18.1 [12.1 to 25.6]
  Swelling: Mild | 17.5 [11.6 to 24.7] | 11.7 [6.5 to 18.8] | 13.8 [8.5 to 20.7]
  Swelling: Moderate | 4.2 [1.6 to 8.9] | 2.5 [0.5 to 7.1] | 3.6 [1.2 to 8.3]
  Swelling: Severe | 0 [0.0 to 2.5] | 0 [0.0 to 3.0] | 0.7 [0.0 to 4.0]
  Pain at Injection Site: Any | 39.9 [31.8 to 48.4] | 22.5 [15.4 to 31.0] | 35.5 [27.6 to 44.1]
  Pain at Injection Site: Mild | 23.8 [17.1 to 31.6] | 17.5 [11.2 to 25.5] | 18.8 [12.7 to 26.4]
  Pain at Injection Site: Moderate | 15.4 [9.9 to 22.4] | 5.0 [1.9 to 10.6] | 15.2 [9.7 to 22.3]
  Pain at Injection Site: Severe | 0.7 [0.0 to 3.8] | 0 [0.0 to 3.0] | 1.4 [0.2 to 5.1]

4. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Dose 4
Description: as for outcome 2
Time Frame: Within 7 Days After Dose 4
Population: The overall safety population included all participants who received at least 1 dose of c7vPnC (in Groups 1 and 2) or Prevnar 13 (in Group 3) and had safety data reported in the study. Here, "Overall Number of Participants Analyzed" signifies number of participants with any e-diary data reported after vaccination in the overall safety population. Dose 4 was fourth dose of c7vPnC in Group 1 and Group 2, and fourth dose of Prevnar 13 in Group 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 105 | 79 | 98
Percentage of participants
  Redness: Any | 22.9 [15.2 to 32.1] | 19.0 [11.0 to 29.4] | 22.4 [14.6 to 32.0]
  Redness: Mild | 21.9 [14.4 to 31.0] | 15.2 [8.1 to 25.0] | 19.4 [12.1 to 28.6]
  Redness: Moderate | 1.0 [0.0 to 5.2] | 3.8 [0.8 to 10.7] | 3.1 [0.6 to 8.7]
  Redness: Severe | 0 [0.0 to 3.5] | 0 [0.0 to 4.6] | 0 [0.0 to 3.7]
  Swelling: Any | 19.0 [12.0 to 27.9] | 13.9 [7.2 to 23.5] | 19.4 [12.1 to 28.6]
  Swelling: Mild | 17.1 [10.5 to 25.7] | 8.9 [3.6 to 17.4] | 13.3 [7.3 to 21.6]
  Swelling: Moderate | 1.9 [0.2 to 6.7] | 5.1 [1.4 to 12.5] | 6.1 [2.3 to 12.9]
  Swelling: Severe | 0 [0.0 to 3.5] | 0 [0.0 to 4.6] | 0 [0.0 to 3.7]
  Pain at Injection Site: Any | 35.2 [26.2 to 45.2] | 22.8 [14.1 to 33.6] | 28.6 [19.9 to 38.6]
  Pain at Injection Site: Mild | 21.9 [14.4 to 31.0] | 16.5 [9.1 to 26.5] | 18.4 [11.3 to 27.5]
  Pain at Injection Site: Moderate | 12.4 [6.8 to 20.2] | 6.3 [2.1 to 14.2] | 10.2 [5.0 to 18.0]
  Pain at Injection Site: Severe | 1.0 [0.0 to 5.2] | 0 [0.0 to 4.6] | 0 [0.0 to 3.7]

5. Primary Outcome: Percentage of Participants With Local Reactions Within 7 Days After Supplemental Dose (SD)
Description: as for outcome 2
Time Frame: Within 7 Days After Supplemental Dose
Population: Participants received Supplemental Dose and had safety data between Supplemental Dose and 1 month after Supplemental Dose. Since supplemental dose was received by participants in reporting arm "Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose", hence data collected and reported for it only and not collected for Group 1 and 2. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 85
Percentage of participants
  Redness: Any | 5.9 [1.9 to 13.2]
  Redness: Mild | 4.7 [1.3 to 11.6]
  Redness: Moderate | 1.2 [0.0 to 6.4]
  Redness: Severe | 0 [0.0 to 4.2]
  Swelling: Any | 9.4 [4.2 to 17.7]
  Swelling: Mild | 9.4 [4.2 to 17.7]
  Swelling: Moderate | 0 [0.0 to 4.2]
  Swelling: Severe | 0 [0.0 to 4.2]
  Pain at Injection Site: Any | 12.9 [6.6 to 22.0]
  Pain at Injection Site: Mild | 11.8 [5.8 to 20.6]
  Pain at Injection Site: Moderate | 1.2 [0.0 to 6.4]
  Pain at Injection Site: Severe | 0 [0.0 to 4.2]

6. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 1
Description: Systemic events were recorded using an e-diary by participant's LAR and included fever, decreased appetite, drowsiness/increased sleep, and irritability. Fever was defined as rectal temperature of greater than or equal to (>=) 38.0 degree Celsius and categorized as >=38.0 to 38.4 degree Celsius,>38.4 to 38.9 degree Celsius, >38.9 to 40.0 degree Celsius and >40.0 degree Celsius. Decreased appetite was graded as mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed). Drowsiness was graded as mild (increased or prolonged sleeping bouts), moderate (slightly subdued, interfered with daily activity) and severe (disabling, not interested in usual daily activity). Irritability: graded as mild (easily consolable), moderate (required increased attention) and severe (inconsolable, crying could not be comforted).
Time Frame: Within 7 Days After Dose 1
Population: The overall safety population included all participants who received at least 1 dose of c7vPnC (in Groups 1 and 2) or Prevnar 13 (in Group 3) and had safety data reported in the study. Here, "Overall Number of Participants Analyzed" signifies number of participants with any e-diary data reported after Dose 1 in overall safety population. Dose 1 was first dose of c7vPnC in Group 1 and Group 2, and first dose of Prevnar 13 in Group 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 166 | 144 | 165
Percentage of participants
  Fever: >=38.0 degree C | 12.7 [8.0 to 18.7] | 5.6 [2.4 to 10.7] | 9.1 [5.2 to 14.6]
  Fever: >=38.0 degree C to 38.4 degree C | 7.8 [4.2 to 13.0] | 3.5 [1.1 to 7.9] | 6.1 [2.9 to 10.9]
  Fever: >38.4 degree C to 38.9 degree C | 3.0 [1.0 to 6.9] | 0.7 [0.0 to 3.8] | 2.4 [0.7 to 6.1]
  Fever: >38.9 degree C to 40.0 degree C | 1.8 [0.4 to 5.2] | 1.4 [0.2 to 4.9] | 0.6 [0.0 to 3.3]
  Fever: >40.0 degree C | 0 [0.0 to 2.2] | 0 [0.0 to 2.5] | 0 [0.0 to 2.2]
  Decreased Appetite: Any | 28.9 [22.2 to 36.4] | 15.3 [9.8 to 22.2] | 26.7 [20.1 to 34.1]
  Decreased Appetite: Mild | 19.3 [13.6 to 26.1] | 6.3 [2.9 to 11.5] | 14.5 [9.5 to 20.9]
  Decreased Appetite: Moderate | 7.2 [3.8 to 12.3] | 9.0 [4.9 to 14.9] | 10.3 [6.1 to 16.0]
  Decreased Appetite: Severe | 2.4 [0.7 to 6.1] | 0 [0.0 to 2.5] | 1.8 [0.4 to 5.2]
  Drowsiness: Any | 59.6 [51.8 to 67.2] | 43.1 [34.8 to 51.6] | 53.3 [45.4 to 61.1]
  Drowsiness: Mild | 41.6 [34.0 to 49.5] | 31.9 [24.4 to 40.2] | 38.2 [30.7 to 46.1]
  Drowsiness: Moderate | 16.3 [11.0 to 22.8] | 9.7 [5.4 to 15.8] | 13.3 [8.5 to 19.5]
  Drowsiness: Severe | 1.8 [0.4 to 5.2] | 1.4 [0.2 to 4.9] | 1.8 [0.4 to 5.2]
  Irritability: Any | 70.5 [62.9 to 77.3] | 57.6 [49.1 to 65.8] | 63.6 [55.8 to 71.0]
  Irritability: Mild | 25.3 [18.9 to 32.6] | 29.2 [21.9 to 37.3] | 23.6 [17.4 to 30.9]
  Irritability: Moderate | 38.0 [30.5 to 45.8] | 23.6 [16.9 to 31.4] | 36.4 [29.0 to 44.2]
  Irritability: Severe | 7.2 [3.8 to 12.3] | 4.9 [2.0 to 9.8] | 3.6 [1.3 to 7.7]

7. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 2
Description: Systemic events were recorded using an e-diary by participant's LAR and included fever, decreased appetite, drowsiness/increased sleep, and irritability. Fever was defined as rectal temperature of >=38.0 degree Celsius and categorized as >=38.0 to 38.4 degree Celsius,>38.4 to 38.9 degree Celsius, >38.9 to 40.0 degree Celsius and >40.0 degree Celsius. Decreased appetite was graded as mild (decreased interest in eating), moderate (decreased oral intake) and severe (refusal to feed). Drowsiness was graded as mild (increased or prolonged sleeping bouts), moderate (slightly subdued, interfered with daily activity) and severe (disabling, not interested in usual daily activity). Irritability: graded as mild (easily consolable), moderate (required increased attention) and severe (inconsolable, crying could not be comforted).
Time Frame: Within 7 Days After Dose 2
Population: The overall safety population included all participants who received at least 1 dose of c7vPnC (in Groups 1 and 2) or Prevnar 13 (in Group 3) and had safety data reported in the study. Here, "Overall Number of Participants Analyzed" signifies number of participants with any e-diary data reported after Dose 2 in overall safety population. Dose 2 was second dose of c7vPnC in Group 1 and Group 2, and second dose of Prevnar 13 in Group 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 152 | 126 | 147
Percentage of participants
  Fever: >=38.0 degree C | 25.7 [18.9 to 33.4] | 4.0 [1.3 to 9.0] | 15.6 [10.2 to 22.5]
  Fever: >=38.0 degree C to 38.4 degree C | 12.5 [7.7 to 18.8] | 3.2 [0.9 to 7.9] | 8.2 [4.3 to 13.8]
  Fever: >38.4 degree C to 38.9 degree C | 10.5 [6.1 to 16.5] | 0.8 [0.0 to 4.3] | 2.7 [0.7 to 6.8]
  Fever: >38.9 degree C to 40.0 degree C | 2.6 [0.7 to 6.6] | 0 [0.0 to 2.9] | 4.1 [1.5 to 8.7]
  Fever: >40.0 degree C | 0 [0.0 to 2.4] | 0 [0.0 to 2.9] | 0.7 [0.0 to 3.7]
  Decreased Appetite: Any | 23.0 [16.6 to 30.5] | 12.7 [7.4 to 19.8] | 25.2 [18.4 to 33.0]
  Decreased Appetite: Mild | 11.8 [7.2 to 18.1] | 8.7 [4.4 to 15.1] | 15.6 [10.2 to 22.5]
  Decreased Appetite: Moderate | 9.9 [5.6 to 15.8] | 4.0 [1.3 to 9.0] | 9.5 [5.3 to 15.5]
  Decreased Appetite: Severe | 1.3 [0.2 to 4.7] | 0 [0.0 to 2.9] | 0 [0.0 to 2.5]
  Drowsiness: Any | 48.7 [40.5 to 56.9] | 21.4 [14.6 to 29.6] | 42.9 [34.7 to 51.3]
  Drowsiness: Mild | 32.2 [24.9 to 40.3] | 15.1 [9.3 to 22.5] | 25.9 [19.0 to 33.7]
  Drowsiness: Moderate | 15.1 [9.8 to 21.8] | 6.3 [2.8 to 12.1] | 17.0 [11.3 to 24.1]
  Drowsiness: Severe | 1.3 [0.2 to 4.7] | 0 [0.0 to 2.9] | 0 [0.0 to 2.5]
  Irritability: Any | 64.5 [56.3 to 72.1] | 44.4 [35.6 to 53.6] | 58.5 [50.1 to 66.6]
  Irritability: Mild | 20.4 [14.3 to 27.7] | 21.4 [14.6 to 29.6] | 17.7 [11.9 to 24.8]
  Irritability: Moderate | 40.8 [32.9 to 49.0] | 20.6 [13.9 to 28.8] | 36.1 [28.3 to 44.4]
  Irritability: Severe | 3.3 [1.1 to 7.5] | 2.4 [0.5 to 6.8] | 4.8 [1.9 to 9.6]

8. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 3
Description: as for outcome 7
Time Frame: Within 7 Days After Dose 3
Population: The overall safety population included all participants who received at least 1 dose of c7vPnC (in Groups 1 and 2) or Prevnar 13 (in Group 3) and had safety data reported in the study. Here, "Overall Number of Participants Analyzed" signifies number of participants with any e-diary data reported after Dose 3 in overall safety population. Dose 3 was third dose of c7vPnC in Group 1 and Group 2, and third dose of Prevnar 13 in Group 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 143 | 120 | 138
Percentage of participants
  Fever: >=38.0 degree C | 14.0 [8.8 to 20.8] | 5.8 [2.4 to 11.6] | 14.5 [9.1 to 21.5]
  Fever: >=38.0 degree C to 38.4 degree C | 6.3 [2.9 to 11.6] | 3.3 [0.9 to 8.3] | 8.0 [4.0 to 13.8]
  Fever: >38.4 degree C to 38.9 degree C | 5.6 [2.4 to 10.7] | 1.7 [0.2 to 5.9] | 2.9 [0.8 to 7.3]
  Fever: >38.9 degree C to 40.0 degree C | 1.4 [0.2 to 5.0] | 0.8 [0.0 to 4.6] | 3.6 [1.2 to 8.3]
  Fever: >40.0 degree C | 0.7 [0.0 to 3.8] | 0 [0.0 to 3.0] | 0 [0.0 to 2.6]
  Decreased Appetite: Any | 19.6 [13.4 to 27.0] | 18.3 [11.9 to 26.4] | 21.0 [14.5 to 28.8]
  Decreased Appetite: Mild | 12.6 [7.6 to 19.2] | 12.5 [7.2 to 19.8] | 10.1 [5.7 to 16.4]
  Decreased Appetite: Moderate | 7.0 [3.4 to 12.5] | 5.8 [2.4 to 11.6] | 10.1 [5.7 to 16.4]
  Decreased Appetite: Severe | 0 [0.0 to 2.5] | 0 [0.0 to 3.0] | 0.7 [0.0 to 4.0]
  Drowsiness: Any | 43.4 [35.1 to 51.9] | 21.7 [14.7 to 30.1] | 45.7 [37.2 to 54.3]
  Drowsiness: Mild | 29.4 [22.1 to 37.6] | 16.7 [10.5 to 24.6] | 32.6 [24.9 to 41.1]
  Drowsiness: Moderate | 13.3 [8.2 to 20.0] | 3.3 [0.9 to 8.3] | 12.3 [7.3 to 19.0]
  Drowsiness: Severe | 0.7 [0.0 to 3.8] | 1.7 [0.2 to 5.9] | 0.7 [0.0 to 4.0]
  Irritability: Any | 57.3 [48.8 to 65.6] | 50.8 [41.6 to 60.1] | 53.6 [44.9 to 62.1]
  Irritability: Mild | 25.2 [18.3 to 33.1] | 26.7 [19.0 to 35.5] | 23.9 [17.1 to 31.9]
  Irritability: Moderate | 31.5 [24.0 to 39.8] | 21.7 [14.7 to 30.1] | 26.8 [19.6 to 35.0]
  Irritability: Severe | 0.7 [0.0 to 3.8] | 2.5 [0.5 to 7.1] | 2.9 [0.8 to 7.3]

9. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Dose 4
Description: as for outcome 7
Time Frame: Within 7 Days After Dose 4
Population: The overall safety population included all participants who received at least 1 dose of c7vPnC (in Groups 1 and 2) or Prevnar 13 (in Group 3) and had safety data reported in the study. Here, "Overall Number of Participants Analyzed" signifies number of participants with any e-diary data reported after Dose 4 in overall safety population. Dose 4 was fourth dose of c7vPnC in Group 1 and Group 2, and fourth dose of Prevnar 13 in Group 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 105 | 79 | 98
Percentage of participants
  Fever: >=38.0 degree C | 12.4 [6.8 to 20.2] | 0 [0.0 to 4.6] | 11.2 [5.7 to 19.2]
  Fever: >=38.0 degree C to 38.4 degree C | 7.6 [3.3 to 14.5] | 0 [0.0 to 4.6] | 4.1 [1.1 to 10.1]
  Fever: >38.4 degree C to 38.9 degree C | 1.9 [0.2 to 6.7] | 0 [0.0 to 4.6] | 4.1 [1.1 to 10.1]
  Fever: >38.9 degree C to 40.0 degree C | 1.9 [0.2 to 6.7] | 0 [0.0 to 4.6] | 3.1 [0.6 to 8.7]
  Fever: >40.0 degree C | 1.0 [0.0 to 5.2] | 0 [0.0 to 4.6] | 0 [0.0 to 3.7]
  Decreased Appetite: Any | 20.0 [12.8 to 28.9] | 13.9 [7.2 to 23.5] | 23.5 [15.5 to 33.1]
  Decreased Appetite: Mild | 14.3 [8.2 to 22.5] | 10.1 [4.5 to 19.0] | 13.3 [7.3 to 21.6]
  Decreased Appetite: Moderate | 4.8 [1.6 to 10.8] | 3.8 [0.8 to 10.7] | 9.2 [4.3 to 16.7]
  Decreased Appetite: Severe | 1.0 [0.0 to 5.2] | 0 [0.0 to 4.6] | 1.0 [0.0 to 5.6]
  Drowsiness: Any | 33.3 [24.4 to 43.2] | 20.3 [12.0 to 30.8] | 29.6 [20.8 to 39.7]
  Drowsiness: Mild | 25.7 [17.7 to 35.2] | 17.7 [10.0 to 27.9] | 20.4 [12.9 to 29.7]
  Drowsiness: Moderate | 7.6 [3.3 to 14.5] | 2.5 [0.3 to 8.8] | 8.2 [3.6 to 15.5]
  Drowsiness: Severe | 0 [0.0 to 3.5] | 0 [0.0 to 4.6] | 1.0 [0.0 to 5.6]
  Irritability: Any | 60.0 [50.0 to 69.4] | 53.2 [41.6 to 64.5] | 46.9 [36.8 to 57.3]
  Irritability: Mild | 24.8 [16.9 to 34.1] | 31.6 [21.6 to 43.1] | 21.4 [13.8 to 30.9]
  Irritability: Moderate | 34.3 [25.3 to 44.2] | 20.3 [12.0 to 30.8] | 23.5 [15.5 to 33.1]
  Irritability: Severe | 1.0 [0.0 to 5.2] | 1.3 [0.0 to 6.9] | 2.0 [0.2 to 7.2]

10. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Supplemental Dose
Description: as for outcome 7
Time Frame: Within 7 Days After Supplemental Dose
Population: Supplemental dose safety analysis set included participants who received Supplemental Dose and had safety data between Supplemental Dose and 1 month after Supplemental Dose. Since supplemental dose was received by participants in reporting arm "Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose", hence data collected and reported for it only and not collected for Group 1 and 2. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 85
Percentage of participants
  Fever: >=38.0 degree C | 5.9 [1.9 to 13.2]
  Fever: >=38.0 degree C to 38.4 degree C | 3.5 [0.7 to 10.0]
  Fever: >38.4 degree C to 38.9 degree C | 1.2 [0.0 to 6.4]
  Fever: >38.9 degree C to 40.0 degree C | 1.2 [0.0 to 6.4]
  Fever: >40.0 degree C | 0 [0.0 to 4.2]
  Decreased Appetite: Any | 11.8 [5.8 to 20.6]
  Decreased Appetite: Mild | 8.2 [3.4 to 16.2]
  Decreased Appetite: Moderate | 1.2 [0.0 to 6.4]
  Decreased Appetite: Severe | 2.4 [0.3 to 8.2]
  Drowsiness: Any | 21.2 [13.1 to 31.4]
  Drowsiness: Mild | 17.6 [10.2 to 27.4]
  Drowsiness: Moderate | 2.4 [0.3 to 8.2]
  Drowsiness: Severe | 1.2 [0.0 to 6.4]
  Irritability: Any | 30.6 [21.0 to 41.5]
  Irritability: Mild | 15.3 [8.4 to 24.7]
  Irritability: Moderate | 12.9 [6.6 to 22.0]
  Irritability: Severe | 2.4 [0.3 to 8.2]

11. Primary Outcome: Percentage of Participants With Adverse Events (AEs) From Dose 1 to 1 Month After Dose 3
Description: An AE was any untoward medical occurrence in study participants who received study vaccine without regard to possibility of causal relationship with the treatment.
Time Frame: From Dose 1 to 1 Month After Dose 3 (up to duration of 5 months)
Population: The overall safety population included all participants who received at least 1 dose of c7vPnC (in Groups 1 and 2) or Prevnar 13 (in Group 3) and had safety data reported in the study. Dose 1 was first dose of c7vPnC in Group 1 and Group 2, and first dose of Prevnar 13 in Group 3. Dose 3 was third dose of c7vPnC in Group 1 and Group 2, and third dose of Prevnar 13 in Group 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 171 | 147 | 166
Percentage of participants | 57.9 [50.1 to 65.4] | 65.3 [57.0 to 73.0] | 56.6 [48.7 to 64.3]

12. Primary Outcome: Percentage of Participants With Adverse Events (AEs) From Dose 4 to 1 Month After Dose 4
Description: as for outcome 11
Time Frame: From Dose 4 to 1 Month After Dose 4 (up to duration of 1 month)
Population: Dose 4 safety analysis set included participants who received Dose 4 and had safety data between Dose 4 and 1 month after Dose 4 for Groups 1 and 2 and had safety data between Dose 4 and Supplemental Dose for Group 3. Dose 4 was fourth dose of c7vPnC in Group 1 and Group 2, and fourth dose of Prevnar 13 in Group 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 110 | 85 | 101
Percentage of participants | 23.6 [16.1 to 32.7] | 15.3 [8.4 to 24.7] | 25.7 [17.6 to 35.4]

13. Primary Outcome: Percentage of Participants With Adverse Events (AEs) From Supplemental Dose to 1 Month After Supplemental Dose
Description: as for outcome 11
Time Frame: From Supplemental Dose to 1 Month After Supplemental Dose (up to duration of 1 month)
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 88
Percentage of participants | 18.2 [10.8 to 27.8]

14. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) From Dose 1 to End of the Study
Description: An SAE was any untoward medical occurrence at any dose that resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital anomaly/birth defect or that was considered to be an important medical event.
Time Frame: From Dose 1 to End of the Study (up to duration of 17 months)
Population: The overall safety population included all participants who received at least 1 dose of c7vPnC (in Groups 1 and 2) or Prevnar 13 (in Group 3) and had safety data reported in the study. Dose 1 was first dose of c7vPnC in Group 1 and Group 2, and first dose of Prevnar 13 in Group 3.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 171 | 147 | 166
Percentage of participants | 4.1 [1.7 to 8.3] | 2.7 [0.7 to 6.8] | 5.4 [2.5 to 10.0]

15. Primary Outcome: Percentage of Participants With Newly Diagnosed Chronic Medical Conditions (NDCMCs) From Dose 1 to End of the Study
Description: An NDCMC was defined as a disease or medical condition, not previously identified, that was expected to be persistent or was otherwise long lasting in its effects.
Time Frame: From Dose 1 to End of the Study (up to duration of 17 months)
Population: as for outcome 14
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 171 | 147 | 166
Percentage of participants | 7.6 [4.1 to 12.6] | 3.4 [1.1 to 7.8] | 7.2 [3.8 to 12.3]

16. Secondary Outcome: Pneumococcal Serotype-specific Immunoglobulin G (IgG) Geometric Mean Concentration (GMC) 1 Month After Dose 3
Description: IgG GMCs were determined for each of 7 pneumococcal serotypes (8, 10A, 11A, 12F, 15B, 22F, and 33F) at 1 month after Dose 3. Dose 3 was third dose of c7vPnC in Group 1 and Group 2, and third dose of Prevnar 13 in Group 3.
Time Frame: 1 Month After Dose 3
Population: Dose 3 evaluable immunogenicity population: included all eligible participants, who were randomly assigned to receive the vaccine, aged 42-98 days on the day of Dose 1 for Groups 1 and 3 or aged 63 to 133 days on the day of Dose 1 for Group 2, received 3 doses of assigned vaccine, had valid determinate IgG concentration for at least 1 serotype from 1 month after Dose 3 visit, had blood collection within 27-56 days, inclusive, after Dose 3, and had no major protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 128 | 107 | 109
microgram per milliliter
  Serotype 8 | 2.90 [2.47 to 3.39] | 5.14 [4.41 to 5.99] | 0.03 [0.03 to 0.04]
  Serotype 10A | 2.55 [1.95 to 3.34] | 4.52 [3.59 to 5.69] | 0.03 [0.03 to 0.04]
  Serotype 11A | 4.37 [3.57 to 5.34] | 8.88 [7.25 to 10.87] | 0.01 [0.01 to 0.02]
  Serotype 12F | 1.92 [1.58 to 2.34] | 3.35 [2.75 to 4.07] | 0.02 [0.02 to 0.02]
  Serotype 15B | 9.12 [7.54 to 11.04] | 14.86 [12.65 to 17.44] | 0.05 [0.04 to 0.06]
  Serotype 22F | 9.25 [7.50 to 11.41] | 23.94 [19.88 to 28.82] | 0.01 [0.01 to 0.01]
  Serotype 33F | 3.40 [2.75 to 4.21] | 4.83 [3.99 to 5.84] | 0.06 [0.05 to 0.06]

17. Secondary Outcome: Percentage of Participants Achieving Prespecified Level of Pneumococcal Serotype-specific Immunoglobulin G (IgG) Concentrations 1 Month After Dose 3
Description: Percentage of participants with pre-specified IgG concentration (>=0.35 microgram per milliliter) were determined for each of 7 pneumococcal serotypes (8, 10A, 11A, 12F, 15B, 22F, and 33F) at 1 month after Dose 3. Dose 3 was third dose of c7vPnC in Group 1 and Group 2, and third dose of Prevnar 13 in Group 3.
Time Frame: 1 Month after Dose 3
Population: as for outcome 16
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 128 | 107 | 109
Percentage of participants
  Serotype 8 | 98.4 [94.5 to 99.8] | 100.0 [96.6 to 100.0] | 1.8 [0.2 to 6.5]
  Serotype 10A | 89.8 [83.3 to 94.5] | 98.1 [93.4 to 99.8] | 2.8 [0.6 to 7.8]
  Serotype 11A | 96.9 [92.2 to 99.1] | 99.1 [94.9 to 100.0] | 0.9 [0.0 to 5.0]
  Serotype 12F | 95.3 [90.1 to 98.3] | 98.1 [93.4 to 99.8] | 0.0 [0.0 to 3.3]
  Serotype 15B | 96.9 [92.2 to 99.1] | 100.0 [96.6 to 100.0] | 6.4 [2.6 to 12.8]
  Serotype 22F | 96.9 [92.2 to 99.1] | 100.0 [96.6 to 100.0] | 0.0 [0.0 to 3.3]
  Serotype 33F | 96.1 [91.1 to 98.7] | 99.1 [94.9 to 100.0] | 4.6 [1.5 to 10.4]

18. Secondary Outcome: Pneumococcal Serotype-specific Immunoglobulin G (IgG) Geometric Mean Concentration (GMC) 1 Month After Dose 4
Description: IgG GMCs were determined for each of 7 pneumococcal serotypes (8, 10A, 11A, 12F, 15B, 22F, and 33F ) at 1 month after Dose 4. Dose 4 was fourth dose of c7vPnC in Group 1 and Group 2, and fourth dose of Prevnar 13 in Group 3.
Time Frame: 1 Month After Dose 4
Population: Dose 4 evaluable immunogenicity population: eligible participants, randomly assigned to receive vaccine, aged 42-98 days on the day of Dose 1 for Groups 1 and 3 or aged 63 to 133 days on the day of Dose 1 for Group 2, received all 4 doses of assigned vaccine, with Dose 4 received in defined window (365-386 days of age), had valid determinate IgG concentration for at least 1 serotype 1 month post dose 4,had blood collection within 27-56 days post Dose 4, and had no major protocol deviations.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
Number analyzed (Participants) | 76 | 57 | 68
microgram per milliliter
  Serotype 8 | 3.79 [3.10 to 4.62] | 3.05 [2.46 to 3.78] | 0.08 [0.06 to 0.12]
  Serotype 10A | 12.77 [10.16 to 16.06] | 7.15 [5.26 to 9.72] | 0.04 [0.03 to 0.04]
  Serotype 11A | 8.25 [6.72 to 10.12] | 7.12 [5.53 to 9.15] | 0.02 [0.01 to 0.04]
  Serotype 12F | 3.15 [2.64 to 3.74] | 2.57 [2.08 to 3.19] | 0.03 [0.02 to 0.03]
  Serotype 15B | 24.56 [21.23 to 28.41] | 17.70 [14.31 to 21.89] | 0.06 [0.04 to 0.07]
  Serotype 22F | 25.68 [21.33 to 30.91] | 29.92 [24.21 to 36.98] | 0.01 [0.01 to 0.02]
  Serotype 33F | 5.38 [4.47 to 6.48] | 3.95 [3.16 to 4.93] | 0.06 [0.05 to 0.08]

ADVERSE EVENTS:
Time Frame: Local reactions, systemic events: within 7 days after Dose 1, 2, 3, 4, Supplemental Dose; Non-SAEs: from Dose 1 to 1 month after Dose 3, Dose 4 to 1 month after Dose 4, Supplemental Dose to 1 month after Supplemental Dose ; SAEs: Dose 1 to 6 months after last dose (Dose 4 or Supplemental Dose) (up to duration of 17 months)
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Overall safety analysis set was analyzed.
Arm/Group | Group 1: c7vPnC and Prevnar 13 Co-administration | Group 2: c7vPnC and Prevnar 13 Staggered Administration | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose
All-Cause Mortality (participants affected / at risk) | 0/171 | 0/147 | 0/166
Serious Adverse Events (participants affected / at risk) | 7/171 | 4/147 | 9/166
Other Adverse Events (participants affected / at risk) | 163/171 | 138/147 | 163/166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: c7vPnC and Prevnar 13 Co-administration (N=171) | Group 2: c7vPnC and Prevnar 13 Staggered Administration (N=147) | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose (N=166)
Bronchiolitis (Infections and infestations) | 2 | 1 | 3
Cellulitis (Infections and infestations) | 0 | 1 | 0
Parotid abscess (Infections and infestations) | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 2
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0
Febrile convulsion (Nervous system disorders) | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 1 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: c7vPnC and Prevnar 13 Co-administration (N=171) | Group 2: c7vPnC and Prevnar 13 Staggered Administration (N=147) | Group 3: Prevnar 13 as Control With Supplemental c7vPnC Dose (N=166)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 2 | 2
Craniosynostosis (Congenital, familial and genetic disorders) | 0 | 2 | 0
Plagiocephaly (Congenital, familial and genetic disorders) | 0 | 0 | 4
Cerumen impaction (Ear and labyrinth disorders) | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 8 | 8 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 6 | 8
Gastritis (Gastrointestinal disorders) | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 2 | 4
Teething (Gastrointestinal disorders) | 4 | 0 | 5
Vomiting (Gastrointestinal disorders) | 5 | 1 | 5
Injection site erythema (REDNESS) (General disorders) | 82 | 67 | 77
Injection site pain (PAIN) (General disorders) | 131 | 82 | 112
Injection site swelling (SWELLING) (General disorders) | 74 | 49 | 68
Pyrexia (General disorders) | 5 | 8 | 7
Pyrexia (FEVER) (General disorders) | 62 | 20 | 53
Food allergy (Immune system disorders) | 2 | 0 | 0
Hypersensitivity (Immune system disorders) | 3 | 0 | 0
Milk allergy (Immune system disorders) | 2 | 0 | 0
Seasonal allergy (Immune system disorders) | 2 | 0 | 2
Acute sinusitis (Infections and infestations) | 2 | 0 | 2
Body tinea (Infections and infestations) | 2 | 1 | 2
Bronchiolitis (Infections and infestations) | 13 | 6 | 14
Bronchitis (Infections and infestations) | 5 | 7 | 3
Candida infection (Infections and infestations) | 0 | 2 | 3
Conjunctivitis (Infections and infestations) | 13 | 8 | 11
Conjunctivitis bacterial (Infections and infestations) | 2 | 1 | 4
Croup infectious (Infections and infestations) | 3 | 2 | 5
Exanthema subitum (Infections and infestations) | 2 | 2 | 0
Gastroenteritis (Infections and infestations) | 2 | 2 | 3
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 2
Hand-foot-and-mouth disease (Infections and infestations) | 3 | 0 | 2
Impetigo (Infections and infestations) | 0 | 2 | 1
Influenza (Infections and infestations) | 3 | 7 | 5
Laryngitis (Infections and infestations) | 0 | 4 | 0
Nasopharyngitis (Infections and infestations) | 4 | 1 | 3
Oral candidiasis (Infections and infestations) | 2 | 3 | 2
Otitis media (Infections and infestations) | 11 | 17 | 13
Otitis media acute (Infections and infestations) | 6 | 2 | 6
Pharyngitis (Infections and infestations) | 4 | 6 | 4
Pneumonia (Infections and infestations) | 1 | 1 | 2
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1 | 3
Respiratory syncytial virus infection (Infections and infestations) | 1 | 2 | 1
Respiratory tract infection viral (Infections and infestations) | 1 | 2 | 1
Roseola (Infections and infestations) | 0 | 0 | 2
Sinusitis (Infections and infestations) | 1 | 3 | 0
Tonsillitis (Infections and infestations) | 3 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 45 | 43 | 35
Urinary tract infection (Infections and infestations) | 3 | 1 | 0
Viral infection (Infections and infestations) | 5 | 4 | 7
Viral upper respiratory tract infection (Infections and infestations) | 4 | 4 | 4
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 2 | 2
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 2 | 3 | 0
Decreased appetite (DECREASED APPETITE) (Metabolism and nutrition disorders) | 82 | 51 | 84
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Somnolence (DROWSINESS) (Nervous system disorders) | 124 | 80 | 126
Irritability (IRRITABILITY) (Psychiatric disorders) | 141 | 113 | 141
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 4
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 4 | 10
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 5 | 5
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 3
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 11 | 5 | 12
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 11 | 7 | 5
Eczema (Skin and subcutaneous tissue disorders) | 5 | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 4 | 1 | 2
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 0 | 3
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/13/NCT03550313/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/13/NCT03550313/SAP_001.pdf